CLINICAL TRIAL: NCT01322854
Title: Randomized Phase III Trial Comparing Intensity Modulated Radiotherapy With Integrated Boost to Conventional Radiotherapy With Consecutive Boost in Patients With Breast Cancer After Breast Conserving Surgery
Brief Title: Adjuvant Whole Breast Radiotherapy (RT) With Intensity Modulated Radiotherapy (IMRT) and a Simultaneous Integrated Boost Versus Conventional RT and a Sequential Boost
Acronym: IMRT-MC2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: DLR German Aerospace Center (Other)
Responsible Party: Juergen Debus, Prof. Dr. Dr., University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMRT-MC2
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer
Keywords: IMRT; Integrated boost; adjuvant radiotherapy; breast cancer; breast conserving surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMRT + integrated boost (Experimental): 28 fractions delivering 50.4 Gy to the whole breast and 64.4 Gy to the tumor-bed by an integrated boost
  Interventions: Radiation: IMRT with an simultaneous integrated boost
- Conventional RT + sequential boost (Other): Conventional radiotherapy of the whole breast in 28 fractions to a dose of 50.4 Gy and a consecutive boost in 8 fractions to a total dose of 66.4 Gy
  Interventions: Radiation: IMRT with an simultaneous integrated boost

INTERVENTIONS:
Radiation: IMRT with an simultaneous integrated boost — IMRT in 28 fractions delivering 50.4 Gy to the whole breast and 64.4 Gy to the tumor-bed

SUMMARY:
The IMRT-MC2 study is a prospective, two armed, multicenter, randomized phase-III-trial comparing intensity modulated radiotherapy with integrated boost to conventional radiotherapy with consecutive boost in patients with breast cancer after breast conserving surgery. 502 patients will be recruited and randomized in two arms: patients in arm A will receive IMRT in 28 fractions delivering 50.4 Gy to the breast and 64.4 Gy to the tumor-bed by an integrated boost, while patients in arm B will receive conventional radiotherapy of the breast in 28 fractions to a dose of 50.4 Gy and a consecutive boost in 8 fractions to a total dose of 66.4 Gy. Primary aim of the study is the assessment of the cosmetic outcome and local control after breast radiotherapy. The study hypothesis is that intensity modulated radiotherapy (IMRT) is, in spite of the reduced treatment duration, at least equivalent to conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years and < 70 years after breast conserving surgery.
* Patients aged ≥ 70 years with following risk factors:

  * Tumor stadium ≥ T2
  * Multifocal disease
  * Lymphangiosis
  * Extended intraductal component
  * Resection margin ≤3mm

Exclusion Criteria:

* Refusal of the patients to be included in the study
* Karnofsky Performance Score ≤ 70%
* Metastatic disease (M1)
* Other malignancies
* Previous radiotherapy of the breast
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
cosmetic results | 2 years
  The cosmetic outcome will be assessed by two independent investigators using the Harvard criteria (excellent, good, fair, poor). Additional parameters to be evaluated are skin color, teleangiectasy, scars, shrinking and asymmetry. Evaluation will also be carried out using a quantitative digitizer scoring system based on standardized photodocumentations of the breast, as described by Vrieling et al.. by calculation of a breast retraction assessment (BRA) score.
local recurrence rates | 5 years

SECONDARY OUTCOMES:
fraction of patients surviving (overall survival) | 15 years
  ratio of number of patients alive to total number of patients treated
fraction of patients surviving without tumor recurrence (disease-free survival) | 15 years
  ratio of patients alive without tumor recurrence to total number of patients treated
quality of life | 2 years
  EORTC questionnaires QLQ-C30 and QLQ-BR23
occurence of secondary malignancies | 15 years
  ratio of patients with occurence of secondary malignancies to total number of patients treated

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, MD, PhD, Principal Investigator — Heidelberg University
Locations (2):
- Germany (2):
  - University of Heidelberg, Dept. Radiation Oncology, Heidelberg
  - University of Heidelberg, Dept. Radiation Oncology, Mannheim

REFERENCES:
- [Derived] Forster T, Hommertgen A, Hafner MF, Arians N, Konig L, Harrabi SB, Schlampp I, Kohler C, Meixner E, Heinrich V, Weidner N, Husing J, Sohn C, Heil J, Golatta M, Hof H, Krug D, Debus J, Horner-Rieber J. Quality of life after simultaneously integrated boost with intensity-modulated versus conventional radiotherapy with sequential boost for adjuvant treatment of breast cancer: 2-year results of the multicenter randomized IMRT-MC2 trial. Radiother Oncol. 2021 Oct;163:165-176. doi: 10.1016/j.radonc.2021.08.019. Epub 2021 Sep 1. PMID 34480960
- [Derived] Horner-Rieber J, Forster T, Hommertgen A, Haefner MF, Arians N, Konig L, Harrabi SB, Schlampp I, Weykamp F, Lischalk JW, Heinrich V, Weidner N, Husing J, Sohn C, Heil J, Hof H, Krug D, Debus J. Intensity Modulated Radiation Therapy (IMRT) With Simultaneously Integrated Boost Shortens Treatment Time and Is Noninferior to Conventional Radiation Therapy Followed by Sequential Boost in Adjuvant Breast Cancer Treatment: Results of a Large Randomized Phase III Trial (IMRT-MC2 Trial). Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1311-1324. doi: 10.1016/j.ijrobp.2020.12.005. Epub 2020 Dec 13. PMID 33321192
- [Derived] Krug D, Koder C, Hafner MF, Arians N, Harrabi SB, Koerber SA, Forster T, Schlampp I, Sohn C, Heil J, Hof H, Horner-Rieber J, Debus J. Acute toxicity of normofractionated intensity modulated radiotherapy with simultaneous integrated boost compared to three-dimensional conformal radiotherapy with sequential boost in the adjuvant treatment of breast cancer. Radiat Oncol. 2020 Oct 13;15(1):235. doi: 10.1186/s13014-020-01652-x. PMID 33050920
- [Derived] Askoxylakis V, Jensen AD, Hafner MF, Fetzner L, Sterzing F, Heil J, Sohn C, Husing J, Tiefenbacher U, Wenz F, Debus J, Hof H. Simultaneous integrated boost for adjuvant treatment of breast cancer--intensity modulated vs. conventional radiotherapy: the IMRT-MC2 trial. BMC Cancer. 2011 Jun 15;11:249. doi: 10.1186/1471-2407-11-249. PMID 21676232